CLINICAL TRIAL: NCT02043132
Title: Intravenous Tranexamic Acid to Reduce Blood Loss in Reverse Total Shoulder Arthroplasty
Brief Title: Tranexamic Acid in Reverse Total Shoulder Arthroplasty
Acronym: TXA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Michael Wiater, MD, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-060
Record Dates: First submitted 2014-01-15; First posted 2014-01-23 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Shoulder Joint Disease; Complications; Arthroplasty; Intraoperative Complications; Blood Loss, Surgical
Keywords: reverse shoulder arthroplasty; Rotator cuff; Orthopedic joint surgery; Total shoulder; Perioperative bleeding; Tranexamic acid; Orthopedic complications; Hemorrhage; Postoperative Hemorrhage; Pathologic Processes; Arthritis; Joint Diseases; Musculoskeletal Diseases; Postoperative Complications; Antifibrinolytic Agents; Fibrin Modulating Agents; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Hemostatics; Coagulants; Hematologic Agents; Therapeutic Uses
MeSH Terms: conditions — Intraoperative Complications; Blood Loss, Surgical; Hemorrhage; Postoperative Hemorrhage; Pathologic Processes; Arthritis; Joint Diseases; Musculoskeletal Diseases; Postoperative Complications | interventions — Tranexamic Acid; Antifibrinolytic Agents; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): Infusion Tranexamic acid on study subjects. They will be randomized to receive an infusion of the standard dose of Tranexamic acid (10mg/kg) One dose will be given by the bedside nurse within 60 minutes prior to surgery and a second dose will be given at wound closure. Infusion will be given along with standard preoperative and operative infusion; no additional infusion will be necessary.
  Interventions: Drug: Tranexamic Acid
- Normal Saline (Placebo Comparator): Infusion of placebo on study subjects. They will be randomized to receive an infusion of placebo (an equivalent volume of normal saline). One dose will be given by the bedside nurse within 60 minutes prior to surgery and a second dose will be given at wound closure. Infusion will be given along with standard preoperative and operative infusion; no additional infusion will be necessary.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Patients randomized to TXA receive an infusion of the standard dose of Tranexamic acid (10 mg/kg) within 60 minutes prior to surgery and at wound closure. The pharmacy uses the randomization list in sequential order to determine whether that patient will receive Tranexamic acid or placebo and will provide two unlabeled IV bags (patient receives two doses) of the appropriate solution.
  Other Names: TXA; Antifibrinolytic
  Arms: Tranexamic acid
Drug: Placebo — Patients randomized to placebo receive an infusion of 10 mg/kg of normal saline within 60 minutes prior to surgery and at wound closure. The pharmacy uses the randomization list in sequential order to determine whether that patient will receive Tranexamic acid or placebo and will provide two unlabeled IV bags (patient receives two doses) of the appropriate solution.
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
To the Investigators' knowledge, TXA has not been studied in the setting of reverse total shoulder arthroplasty. We propose a double-blinded, randomized, controlled trial comparing perioperative administration of TXA to placebo in the setting of RTSA. The purpose of this study is to examine the efficacy of TXA in reducing overall blood loss and transfusion rates in patients undergoing reverse total shoulder arthroplasty.

DETAILED DESCRIPTION:
Shoulder arthroplasty is a procedure used to relieve pain and dysfunction associated with arthritic destruction of the gleno-humeral joint. It has been demonstrated that in patients with concomitant rotator cuff deficiency, reverse total shoulder arthroplasty (rTSA) is an efficacious procedure that relieves pain as well as increases the lever-arm of the deltoid muscle, thus improving post-operative strength and range of motion.

However, perioperative blood loss in total shoulder arthroplasty can be significant, with an overall rate of allogeneic blood transfusion reported to be 7.4%-43% [1-5]. Patients undergoing reverse total shoulder arthroplasty are at even further risk of requiring a postoperative blood transfusion [2]. Blood transfusions are associated with significant risks to patient health that range from mild to life threatening.

Tranexamic acid (TXA) is an antifibrinolytic medication (reduces the destruction of blood clots, thus promoting the ability to stop bleeding) that is frequently used to reduce perioperative blood loss, blood transfusions and associated costs in major cardiac, vascular, obstetric, and orthopedic procedures. Currently, TXA is increasingly used in orthopedic joint reconstructive surgery and has proven to be safe and effective in reducing blood loss following total knee arthroplasty (TKA) and total hip arthroplasty (THA) [11-33]. Multiple recent meta-analyses have found that use of TXA in the setting of TKA and THA leads to significantly less overall blood loss and lower rates of blood transfusion without increasing rates of venous thromboembolism (VTE) or other complications [34-37]. TXA is now on formulary at William Beaumont Hospital.

100 patients slated to undergo elective reverse total shoulder arthroplasty will be recruited and randomized to receive either an infusion of the standard dose of TXA (10mg/kg) or placebo (an equivalent volume of normal saline) within 60 minutes prior to surgery and at wound closure.

Adult subjects 18 years of age or older will participate in this study after the objectives, methods, and potential hazards of the study have been fully explained, and after they have signed the informed consent form. The Investigator or designee is responsible for keeping a record of all subjects who sign an informed consent form for entry into this study

DATA AND SAFETY MONITORING PLAN Beaumont Research will follow their standard operating policy and procedure for establishing a group of designated Beaumont Hospital faculty that will be responsible for data and safety monitoring. This group will include a clinician, physician, scientific member and statistician. They will meet twice throughout the course of the study. A medical monitor was not appointed since this is a single-site study; Dr. J. Michael Wiater will personally oversee the health and well-being of all patients and submit AE reports, and the designated group will directly review all adverse event reports. Beaumont's Human Investigation Committee will review the data safety monitoring plan as part of their IRB approval process.

Study data will be transcribed by study personnel from the source documents into an electronic database maintained in Excel. The data collections forms are to be completed by the research nurse at the time of the data collection so that they always reflect the latest observations on the subjects participating in the study. Demographic data will be filled in preoperatively, intraoperative blood loss will be recorded in the OR, postoperative blood loss and transfusion will be collected retrospectively, and complications will be recorded as they occur or at 2 and 6 week follow-up. All data entries, corrections and alterations must be made by the investigator or other authorized study personnel. The Research Institute will complete internal auditing at random intervals during the study for data integrity, proper informed consent process implementation and documentation, protocol adherence, and patient safety reporting compliance to regulatory bodies.

Descriptive statistics will be provided for all data collected. Missing data will remain missing and will not be replaced by substitutions or interpolations. Statistical software (SPSS, IBM, Inc) will be used for all analyses. Baseline and demographic data will be compared between the 2 randomization arms to determine if any imbalances exist. Categorical variables will be shown as counts and % frequencies. They will be examined using Pearson's Chi-square where appropriate (expected frequency>5), otherwise a Fisher's Exact test will be used. Continuous variables will be examined for normality. Normally distributed variables will be analyzed using t-tests and non-normally distributed variables will be examined using non-parametric Wilcoxon rank tests. All continuous variables will be shown as means+/- the standard deviation followed by the median and (25th, 75th percentiles) where needed.

The primary outcome of intraoperative and postoperative blood loss and postoperative drop in Hb will be examined for normality. Normally distributed variables will be analyzed using t-tests and non-normally distributed variables will be examined using non-parametric Wilcoxon rank tests. Total number of postoperative transfusions and total number of patients requiring postoperative transfusions will be shown as counts and % frequencies. They will be examined using Pearson's Chi-square where appropriate (expected frequency>5), otherwise a Fisher's Exact test will be used.

The secondary outcomes of systemic and surgical site complications will be examined between the two randomization arms using Pearson's Chi-square where appropriate (expected frequency>5), otherwise a Fisher's Exact test will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing scheduled primary reverse total shoulder arthroplasty performed by J. Michael Wiater, MD.
2. Patients age 18 and older

Exclusion Criteria:

1. Pregnant* or breast-feeding women
2. Allergy to tranexamic acid
3. Acquired disturbances of color vision
4. Use of estrogen containing medications (i.e. oral contraceptive pills)
5. Hormone replacement therapy
6. Preoperative anemia [Hemoglobin (Hb) < 11g/dL in females, Hb < 12 g/dL in males]
7. Refusal of blood products
8. Preoperative use of anticoagulant therapy within 5 days prior to surgery

   1. Coumadin
   2. Heparin
   3. Low molecular weight heparin
   4. Factor Xa inhibitors
9. Thrombin inhibitors
10. Coagulopathy
11. Thrombophilia
12. Antithrombin deficiency
13. Factor V Leiden
14. Antiphospholipid Syndrome
15. Protein C and S deficiency
16. History of heparin induced thrombocytopenia
17. Sickle cell anemia
18. Myeloproliferative disorders
19. Platelet < 150,00 mm3
20. International Normalized Ratio (INR) > 1.4
21. Partial Thromboplastin Time (PTT) > 1.4 times normal
22. A history of arterial or venous thromboembolism
23. Cerebral Vascular Accident
24. Deep Vein Thrombosis
25. Pulmonary Embolism
26. Subarachnoid hemorrhage
27. Active intravascular clotting
28. Major comorbidities
29. Coronary artery disease (New York Heart Association Class III or IV)
30. Previous MI
31. Severe pulmonary disease (FEV <50% normal)
32. Plasma creatinine > 115 μmol/L in males, > 100 μmol/L in females, or hepatic failure)

34. Participation in another clinical trial 35. *All women of child bearing potential must have a negative serum or urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Wiater, M.D., Principal Investigator — Corewell Health East; Kevin Baker, PhD, Study Director — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardy JC, Hung M, Snow BJ, Martin CL, Tashjian RZ, Burks RT, Greis PE. Blood transfusion associated with shoulder arthroplasty. J Shoulder Elbow Surg. 2013 Feb;22(2):233-9. doi: 10.1016/j.jse.2012.04.013. Epub 2012 Aug 29. PMID 22938787
- [Background] Gruson KI, Accousti KJ, Parsons BO, Pillai G, Flatow EL. Transfusion after shoulder arthroplasty: an analysis of rates and risk factors. J Shoulder Elbow Surg. 2009 Mar-Apr;18(2):225-30. doi: 10.1016/j.jse.2008.08.005. Epub 2008 Dec 31. PMID 19119020
- [Background] Schumer RA, Chae JS, Markert RJ, Sprott D, Crosby LA. Predicting transfusion in shoulder arthroplasty. J Shoulder Elbow Surg. 2010 Jan;19(1):91-6. doi: 10.1016/j.jse.2009.05.001. PMID 19664937
- [Background] Millett PJ, Porramatikul M, Chen N, Zurakowski D, Warner JJ. Analysis of transfusion predictors in shoulder arthroplasty. J Bone Joint Surg Am. 2006 Jun;88(6):1223-30. doi: 10.2106/JBJS.E.00706. PMID 16757754
- [Background] Sperling JW, Duncan SF, Cofield RH, Schleck CD, Harmsen WS. Incidence and risk factors for blood transfusion in shoulder arthroplasty. J Shoulder Elbow Surg. 2005 Nov-Dec;14(6):599-601. doi: 10.1016/j.jse.2005.03.006. PMID 16337526
- [Background] Samama CM. A direct antifibrinolytic agent in major orthopedic surgery. Orthopedics. 2004 Jun;27(6 Suppl):s675-80. doi: 10.3928/0147-7447-20040602-09. PMID 15239556
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Hardy JF, Desroches J. Natural and synthetic antifibrinolytics in cardiac surgery. Can J Anaesth. 1992 Apr;39(4):353-65. doi: 10.1007/BF03009046. PMID 1373346
- [Background] Burry M. The decerebrate patient. J Neurosurg Nurs. 1979 Mar;11(1):6-9. No abstract available. PMID 255562
- [Background] Prentice CR. Basis of antifibrinolytic therapy. J Clin Pathol Suppl (R Coll Pathol). 1980;14:35-40. No abstract available. PMID 6159375
- [Background] Alvarez JC, Santiveri FX, Ramos I, Vela E, Puig L, Escolano F. Tranexamic acid reduces blood transfusion in total knee arthroplasty even when a blood conservation program is applied. Transfusion. 2008 Mar;48(3):519-25. doi: 10.1111/j.1537-2995.2007.01564.x. Epub 2007 Dec 7. PMID 18067499
- [Background] Benoni G, Fredin H. Fibrinolytic inhibition with tranexamic acid reduces blood loss and blood transfusion after knee arthroplasty: a prospective, randomised, double-blind study of 86 patients. J Bone Joint Surg Br. 1996 May;78(3):434-40. PMID 8636182
- [Background] Camarasa MA, Olle G, Serra-Prat M, Martin A, Sanchez M, Ricos P, Perez A, Opisso L. Efficacy of aminocaproic, tranexamic acids in the control of bleeding during total knee replacement: a randomized clinical trial. Br J Anaesth. 2006 May;96(5):576-82. doi: 10.1093/bja/ael057. Epub 2006 Mar 10. PMID 16531440
- [Background] Ellis MH, Fredman B, Zohar E, Ifrach N, Jedeikin R. The effect of tourniquet application, tranexamic acid, and desmopressin on the procoagulant and fibrinolytic systems during total knee replacement. J Clin Anesth. 2001 Nov;13(7):509-13. doi: 10.1016/s0952-8180(01)00319-1. PMID 11704449
- [Background] Good L, Peterson E, Lisander B. Tranexamic acid decreases external blood loss but not hidden blood loss in total knee replacement. Br J Anaesth. 2003 May;90(5):596-9. doi: 10.1093/bja/aeg111. PMID 12697586
- [Background] Hiippala ST, Strid LJ, Wennerstrand MI, Arvela JV, Niemela HM, Mantyla SK, Kuisma RP, Ylinen JE. Tranexamic acid radically decreases blood loss and transfusions associated with total knee arthroplasty. Anesth Analg. 1997 Apr;84(4):839-44. doi: 10.1097/00000539-199704000-00026. PMID 9085968
- [Background] Jansen AJ, Andreica S, Claeys M, D'Haese J, Camu F, Jochmans K. Use of tranexamic acid for an effective blood conservation strategy after total knee arthroplasty. Br J Anaesth. 1999 Oct;83(4):596-601. doi: 10.1093/bja/83.4.596. PMID 10673876
- [Background] Kakar PN, Gupta N, Govil P, Shah V. Efficacy and Safety of Tranexamic Acid in Control of Bleeding Following TKR: A Randomized Clinical Trial. Indian J Anaesth. 2009 Dec;53(6):667-71. PMID 20640094
- [Background] MacGillivray RG, Tarabichi SB, Hawari MF, Raoof NT. Tranexamic acid to reduce blood loss after bilateral total knee arthroplasty: a prospective, randomized double blind study. J Arthroplasty. 2011 Jan;26(1):24-8. doi: 10.1016/j.arth.2009.11.013. Epub 2010 Feb 19. PMID 20171048
- [Background] Orpen NM, Little C, Walker G, Crawfurd EJ. Tranexamic acid reduces early post-operative blood loss after total knee arthroplasty: a prospective randomised controlled trial of 29 patients. Knee. 2006 Mar;13(2):106-10. doi: 10.1016/j.knee.2005.11.001. Epub 2006 Feb 17. PMID 16487712
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishima T, Ishii S. Timing of the administration of tranexamic acid for maximum reduction in blood loss in arthroplasty of the knee. J Bone Joint Surg Br. 2001 Jul;83(5):702-5. doi: 10.1302/0301-620x.83b5.11745. PMID 11476309
- [Background] Veien M, Sorensen JV, Madsen F, Juelsgaard P. Tranexamic acid given intraoperatively reduces blood loss after total knee replacement: a randomized, controlled study. Acta Anaesthesiol Scand. 2002 Nov;46(10):1206-11. doi: 10.1034/j.1399-6576.2002.461007.x. PMID 12421192
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Zhang F, Gao Z, Yu J. [Clinical comparative studies on effect of tranexamic acid on blood loss associated with total knee arthroplasty]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2007 Dec;21(12):1302-4. Chinese. PMID 18277670
- [Background] Claeys MA, Vermeersch N, Haentjens P. Reduction of blood loss with tranexamic acid in primary total hip replacement surgery. Acta Chir Belg. 2007 Jul-Aug;107(4):397-401. doi: 10.1080/00015458.2007.11680081. PMID 17966532
- [Background] Ido K, Neo M, Asada Y, Kondo K, Morita T, Sakamoto T, Hayashi R, Kuriyama S. Reduction of blood loss using tranexamic acid in total knee and hip arthroplasties. Arch Orthop Trauma Surg. 2000;120(9):518-20. doi: 10.1007/s004029900132. PMID 11011672
- [Background] Niskanen RO, Korkala OL. Tranexamic acid reduces blood loss in cemented hip arthroplasty: a randomized, double-blind study of 39 patients with osteoarthritis. Acta Orthop. 2005 Dec;76(6):829-32. doi: 10.1080/17453670510045444. PMID 16470437
- [Background] Garneti N, Field J. Bone bleeding during total hip arthroplasty after administration of tranexamic acid. J Arthroplasty. 2004 Jun;19(4):488-92. doi: 10.1016/j.arth.2003.12.073. PMID 15188109
- [Background] Benoni G, Fredin H, Knebel R, Nilsson P. Blood conservation with tranexamic acid in total hip arthroplasty: a randomized, double-blind study in 40 primary operations. Acta Orthop Scand. 2001 Oct;72(5):442-8. doi: 10.1080/000164701753532754. PMID 11728069
- [Background] Ekback G, Axelsson K, Ryttberg L, Edlund B, Kjellberg J, Weckstrom J, Carlsson O, Schott U. Tranexamic acid reduces blood loss in total hip replacement surgery. Anesth Analg. 2000 Nov;91(5):1124-30. doi: 10.1097/00000539-200011000-00014. PMID 11049894
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Lemay E, Guay J, Cote C, Roy A. Tranexamic acid reduces the need for allogenic red blood cell transfusions in patients undergoing total hip replacement. Can J Anaesth. 2004 Jan;51(1):31-7. doi: 10.1007/BF03018543. PMID 14709457
- [Background] Yamasaki S, Masuhara K, Fuji T. Tranexamic acid reduces blood loss after cementless total hip arthroplasty-prospective randomized study in 40 cases. Int Orthop. 2004 Apr;28(2):69-73. doi: 10.1007/s00264-003-0511-4. Epub 2003 Oct 10. PMID 15224162
- [Background] Yang ZG, Chen WP, Wu LD. Effectiveness and safety of tranexamic acid in reducing blood loss in total knee arthroplasty: a meta-analysis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1153-9. doi: 10.2106/JBJS.K.00873. PMID 22623147
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Brecher ME, Monk T, Goodnough LT. A standardized method for calculating blood loss. Transfusion. 1997 Oct;37(10):1070-4. doi: 10.1046/j.1537-2995.1997.371098016448.x. PMID 9354828
- [Background] Aderinto J, Brenkel IJ. Pre-operative predictors of the requirement for blood transfusion following total hip replacement. J Bone Joint Surg Br. 2004 Sep;86(7):970-3. doi: 10.1302/0301-620x.86b7.14682. PMID 15446520

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 116 participants were consented; 2 were lost to follow-up and 12 were screen failures. These 14 participants were excluded from the overall data analysis, therefore 102 completed participants were analyzed.
Period: Overall Study
Arm/Group | Tranexamic Acid | Normal Saline
Started | 58 | 58
Completed | 53 | 49
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — screen failures | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Normal Saline | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 66 (9) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 60
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United States | 53 | 49 | 102

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss
Description: Total Blood Loss as calculated according to method as described by Good et al. Total Blood Loss (mL) = 1000 X Hb(loss)/Hb(initial)
Time Frame: Preoperative through Postoperative Days 1 and 2
Measure: Mean (Standard Deviation); unit: Total Blood Loss (mL)
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
Total Blood Loss (mL) | 1122.4 (411.6) | 1472 (475.4)

2. Primary Outcome: Total Hemoglobin Loss
Description: Total hemoglobin loss estimated using the formula for total blood volume described by Nadler et al Hb(loss) = blood volume (L) x [Hb(initial)(g/L) - Hb(final)(g/L)] + Hb(transfused)
Time Frame: Preoperative through Postoperative Days 1 and 2
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
g | 154.6 [138.0 to 171.2] | 200.1 [181.3 to 218.8]

3. Primary Outcome: Total Drain Output
Description: Total Drain Output as measured postoperatively 0-48 hours
Time Frame: 0-48 hours postoperatively
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
mL | 221 [186 to 256] | 372 [324 to 420]

4. Secondary Outcome: Number of Participants Experiencing Pulmonary Embolism
Description: The occurrence of the following systemic and surgical site complications within 6 weeks of surgery will be recorded. Data will be obtained from EMR and from patient at standard of care 2 week and 6 week follow-up appointment.
  Pulmonary Embolism
Time Frame: up to 6-weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Myocardial Infarction
Description: The occurrence of the following systemic and surgical site complications within 6 weeks of surgery will be recorded. Data will be obtained from EMR and from patient at standard of care 2 week and 6 week follow-up appointment.
  Myocardial infarction
Time Frame: up to 6-weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
Participants | 0 | 1

6. Secondary Outcome: Number of Participants Experiencing Deep Vein Thrombosis
Description: The occurrence of the following systemic and surgical site complications within 6 weeks of surgery will be recorded. Data will be obtained from EMR and from patient at standard of care 2 week and 6 week follow-up appointment.
  Deep venous thrombosis
Time Frame: up to 6-weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing Hematoma as a Surgical Site Complication
Description: The occurrence of the following systemic and surgical site complications within 6 weeks of surgery will be recorded. Data will be obtained from EMR and from patient at standard of care 2 week and 6 week follow-up appointment.
  Hematoma
Time Frame: up to 6-weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
Participants | 0 | 0

8. Secondary Outcome: Number of Participants Experiencing Infection as a Surgical Site Complication
Description: The occurrence of the following systemic and surgical site complications within 6 weeks of surgery will be recorded. Data will be obtained from EMR and from patient at standard of care 2 week and 6 week follow-up appointment.
  Infection
Time Frame: up to 6-weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Normal Saline
Number analyzed (Participants) | 53 | 49
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/49
Other Adverse Events (participants affected / at risk) | 1/53 | 1/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=53) | Normal Saline (N=49)
Non-ST elevation myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Non-ST elevation myocardial infarction from acute blood loss anemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=53) | Normal Saline (N=49)
Skin Allergic Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncopal fall (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No